CLINICAL TRIAL: NCT02193529
Title: Weight Loss and Metabolic Surgery Center Min-Sheng General Hospital
Brief Title: Dietary Intake After Laparoscopic Sleeve Gastrectomy -a 5 Year Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Principal Investigator, WEI-CHENG YAO, Institutional Review Board, Min-Sheng General Hospital
Other Study IDs: DIA-LSG; DIA5y (Other: Asia Pacific Bariatric surgery center)
Record Dates: First submitted 2014-07-08; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Morbid Obesity
Keywords: sleeve gastrectomy, dietary intake, morbid obesity.
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Weight reducing surgery is the only effective therapy for morbid obese patients.

Sleeve gastrectomy is a popular choice for bariatric surgery because of less sequela. There is poor knowledge about the nutritional status inpatients after LSG. The aim of our study was to investigate the relationship between dietary intake and weight loss after LSG.

DETAILED DESCRIPTION:
Weight reducing surgery is the only effective therapy for morbid obese patients. Restrictive type surgery is safer than mal-absorptive type surgery. Laparoscopic sleeve gastrectomy is an effective surgery. In laparoscopic sleeve gastrectomy (LSG), about 90% of the stomach is surgically removed by vertical resection of the great curvature side, including the fundus. The simplicity of surgical procedures, the low occurrence of complications, and the efficiency of reducing excess weight have made LSG as a popular choice for bariatric surgery. After LSG, the amount of food eaten is drastically reduced, leading to nutritional deficiencies potentially. There is poor knowledge about the nutritional status inpatients after LSG. Some literatures suggest that LSG results in less nutritional deficiencies than Roux-en-Y gastric bypass. The aim of our study was to investigate the relationship between dietary intake and weight loss after LSG.

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity patients received laparoscopic sleeve gastrectomy for more then 5 years.

BMI above 40 kg/m2 when operation. Age 18-65 years old. No major psychosis or binge eating disorder. No endocrine disease. failed to lose weight with medical therapy.

Exclusion Criteria:

* current hepatitis, under steroid treatment,cancer, thyroid disease,alcoholism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: morbid obesity patients received laparoscopic sleeve gastrectomy for more then 5 years. BMI above 40 kg/m2 when operation. Age 18-65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Dietary intake after laparoscopic sleeve gastrectomy 5 years | up to 18 months
  The aim of this study was to investigate the relationship between dietary intake and weight loss effect after sleeve gastrectomy.The calculation of the majority of the nutrients is based on Australian nutrient composition data. The item include: energy ( kcal/day), protein, fat, carbohydrate, vitamin and minerals.

CONTACTS AND LOCATIONS:
Overall Officials: Ju J Chou, university, Principal Investigator — School of Nutrition and Health Sciences,Taipei Medical University
Locations (1):
- Weight Loss and Metabolic Surgery Center Min-Sheng General Hospital, Taoyuan District, Taoyuan, Taiwan